CLINICAL TRIAL: NCT00043589
Title: Memory and Mental Health in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH035182 (NIH); R01MH035182 (NIH)
Record Dates: First submitted 2002-08-09; First posted 2002-08-13 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Memory Disorders
Keywords: Memory
MeSH Terms: conditions — Memory Disorders | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: donepezil
Procedure: Memory-training class

SUMMARY:
This study will evaluate the effectiveness of donepezil (Aricept®) and cognitive training in improving memory performance in elderly adults.

DETAILED DESCRIPTION:
The drug donepezil plus cognitive training may work better than cognitive training alone to improve the memory of nondemented older adults. In this study, participants are assigned randomly to receive either donepezil plus cognitive training or placebo plus cognitive training. Memory and quality of life tests are used to evaluate the effects of the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental Exam score between 24 and 30
* Hamilton Depression Score of 12 or less on 17-item scale
* Visual and auditory acuity adequate for neuropsychological testing
* General good health (no additional diseases expected to interfere with the study)
* Normal B12, Rapid Plasma Reagin (RPR), and Thyroid Function Tests
* Normal general clinical chemistry, complete blood count, and electrocardiogram (ECG)
* Female participants must be 2 years postmenopausal or surgically sterile

Exclusion Criteria:

* Significant neurologic disease
* Possible or probable Alzheimer's Disease (AD)
* Parkinson's disease
* Multi-infarct dementia
* Huntington's disease
* Normal pressure hydrocephalus
* Brain tumor
* Progressive supranuclear palsy
* Seizure disorder
* Subdural hematoma
* Multiple sclerosis
* History of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities
* Major depression or other major psychiatric disorder as described in DSM IV within the past 2 years
* Psychotic features, agitation, or behavioral problems within the last 3 months
* History of alcohol or substance abuse or dependence within the past 2 years
* Significant systemic illness or unstable medical condition including: a) history of systemic cancer within the last 5 years (nonmetastatic skin cancers are acceptable); b) history of myocardial infarction within the past year or unstable or severe cardiovascular disease, including angina or CHF with symptoms at rest; c) clinically significant obstructive pulmonary disease or asthma; d) clinically significant and unstable gastrointestinal disorder such as ulcer disease or a history of active or occult gastrointestinal bleeding within 2 years; e) clinically significant laboratory test abnormalities on the battery of screening tests (hematology, prothrombin time, chemistry, urinalysis, ECG); f) insulin-requiring diabetes or uncontrolled diabetes mellitus; g) uncontrolled hypertension (systolic BP greater than 170 or diastolic greater than 100); h) history of clinically significant liver disease, coagulopathy, or vitamin K deficiency within the past 2 years
* Use of centrally active beta-blockers, narcotics, methyldopa, and clonidine within 4 weeks prior to screening
* Use of anti-Parkinsonian medications (e.g. Sinemet, amantadine, bromocriptine, pergolide, and selegiline) within 2 months prior to screening
* Use of neuroleptics or narcotic analgesics within 4 weeks prior to screening
* Use of long-acting benzodiazepines or barbiturates within 4 weeks prior to screening
* Use of short-acting anxiolytics or sedative hypnotics more frequently than 2 times per week within 4 weeks prior to screening (note: sedative agents should not be used within 72 hours of screening)
* Initiation or change in dose of an antidepressant lacking significant cholinergic side effects within the 4 weeks prior to screening (use of stable doses of antidepressants for at least 4 weeks prior to screening is acceptable)
* Use of systemic corticosteroids within 3 months prior to screening
* Medications with significant cholinergic or anticholinergic side effects (e.g. pyridostigmine, tricyclic antidepressants, meclizine, and oxybutynin) within 4 weeks prior to screening
* Use of anti-convulsants (e.g. Phenytoin, Phenobarbital, Carbamazepine) within 2 months prior to screening
* Use of warfarin (Coumadin) within 4 weeks prior to screening
* Prior use of any FDA approved medications for the treatment of AD (e.g. tacrine, donepezil, or other newly approved medications)

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-06; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aging Clinical Research Center, VA Palo Alto Health Care System, Palo Alto, California, United States